CLINICAL TRIAL: NCT04584112
Title: A Phase Ib, Open-Label, Multicohort Study of the Safety, Efficacy, and Pharmacokinetics of Tiragolumab in Combination With Atezolizumab and Chemotherapy in Patients With Triple-Negative Breast Cancer
Brief Title: A Study of the Safety, Efficacy, and Pharmacokinetics of Tiragolumab in Combination With Atezolizumab and Chemotherapy in Participants With Triple-Negative Breast Cancer
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CO42177; 2020-000531-47 (EudraCT Number)
Record Dates: First submitted 2020-10-05; First posted 2020-10-12 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Triple-Negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms | interventions — Tiragolumab; atezolizumab; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Carboplatin; Doxorubicin; liposomal doxorubicin; Cyclophosphamide; Granulocyte Colony-Stimulating Factor; Filgrastim; pegfilgrastim; Granulocyte-Macrophage Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Cohort A: Tiragolumab and Atezolizumab + Nab-paclitaxel (Experimental): Participants with first-line metastatic TNBC will receive tiragolumab and atezolizumab on Day 1 of every 28-day cycle plus nab-paclitaxel on Days 1, 8, and 15 of every 28-day cycle.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Nab-paclitaxel
- Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC (Experimental): Participants with early TNBC in the neoadjuvant setting, who are eligible for surgery, will receive tiragolumab and atezolizumab every 2 weeks (Q2W) in combination with nab-paclitaxel weekly (QW) and carboplatin every 3 weeks (Q3W) for four cycles, followed by tiragolumab and atezolizumab in combination with doxorubicin and cyclophosphamide Q2W with granulocyte colony-stimulating factor (G-CSF; filgrastim or pegfilgrastim) or granulocyte-macrophage colony-stimulating factor (GM-CSF) support for four doses.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Nab-paclitaxel; Drug: Carboplatin; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Granulocyte-macrophage colony-stimulating factor (GM-CSF)
- Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC (Experimental): Participantswith early TNBC in the neoadjuvant setting, who are eligible for surgery, will receive tiragolumab and atezolizumab Q2W in combination with nab-paclitaxel QW for 12 weeks, followed by tiragolumab and atezolizumab in combination with doxorubicin and cyclophosphamide Q2W with G-CSF (filgrastim or pegfilgrastim) or GM-CSF support for four doses.
  Interventions: Drug: Tiragolumab; Drug: Atezolizumab; Drug: Nab-paclitaxel; Drug: Doxorubicin; Drug: Cyclophosphamide; Drug: Granulocyte colony-stimulating factor (G-CSF); Drug: Granulocyte-macrophage colony-stimulating factor (GM-CSF)

INTERVENTIONS:
Drug: Tiragolumab — Tiragolumab 840 milligrams (mg) administered by intravenous (IV) infusion on Day 1 of every 28-day cycle.
  Arms: Cohort A: Tiragolumab and Atezolizumab + Nab-paclitaxel
Drug: Atezolizumab — Atezolizumab 1680 mg administered by IV infusion on Day 1 of every 28-day cycle.
  Other Names: Tecentriq
  Arms: Cohort A: Tiragolumab and Atezolizumab + Nab-paclitaxel
Drug: Nab-paclitaxel — Nab-paclitaxel 100 milligrams per square meter (mg/m^2) administered by IV infusion on Days 1, 8, and 15 of every 28-day cycle.
  Other Names: Abraxane
  Arms: Cohort A: Tiragolumab and Atezolizumab + Nab-paclitaxel
Drug: Tiragolumab — Tiragolumab 420 mg administered by IV infusion Q2W.
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Atezolizumab — Atezolizumab 840 mg administered by IV infusion Q2W.
  Other Names: Tecentriq
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Nab-paclitaxel — Nab-paclitaxel 125 mg/m^2 administered by IV infusion QW.
  Other Names: Abraxane
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Carboplatin — Carboplatin (area under the concentration-time curve [AUC]: 5 milligrams per milliliter per minute [mg/mL/min]) administered by IV infusion Q3W.
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Doxorubicin — Doxorubicin 60 mg/m^2 Q2W administered by IV infusion.
  Other Names: Lipodox, Doxil
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Cyclophosphamide — Cyclophosphamide 600 mg/m^2 Q2W administered by IV infusion.
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Granulocyte colony-stimulating factor (G-CSF) — G-CSF support for four doses.
  Other Names: filgrastim, pegfilgrastim
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC
Drug: Granulocyte-macrophage colony-stimulating factor (GM-CSF) — GM-CSF support for four doses.
  Arms: Cohort B: Tiragolumab and Atezolizumab + Nab-pac-AC; Cohort B: Tiragolumab and Atezolizumab + Nab-pac-carbo-AC

SUMMARY:
The purpose of this study is to evaluate the safety, efficacy, and pharmacokinetics of tiragolumab in combination with atezolizumab and chemotherapy in participants with metastatic and early triple-negative breast cancer (TNBC).

ELIGIBILITY:
Inclusion Criteria

Cohort A:

* Metastatic or locally advanced unresectable, histologically documented TNBC characterized by absence of human epidermal growth factor 2 (HER2), estrogen receptor (ER), and progesterone receptor (PR) expression
* Only patients with metastatic TNBC tumors that are centrally tested and found to be programmed death-ligand 1 (PD-L1) positive will be enrolled
* No prior chemotherapy or targeted systemic therapy for inoperable locally advanced or metastatic TNBC
* Eastern Cooperative Oncology Group performance status of 0 or 1
* Measurable disease, as assessed by the investigator according to RECIST v1.1
* Adequate hematologic and end-organ function

Cohort B:

* Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1
* Histologically documented TNBC (negative HER2, ER, and PR status)
* Confirmed tumor PD-L1 evaluation as documented through central testing of a representative tumor tissue specimen
* Primary breast tumor size of greater than (>) 2 centimeters (cm) by at least one radiographic or clinical measurement
* Stage at presentation: cT2-cT4, cN0-cN3, cM0
* Baseline left ventricular ejection fraction (LVEF) greater than or equal to (>/=) 53 percent (%) measured by echocardiogram (ECHO) or multiple-gated acquisition (MUGA) scans
* Adequate hematologic and end-organ function

Exclusion Criteria

Cohort A:

* Formalin-fixed, paraffin-embedded (FFPE) tumor tissue that is PD-L1 negative, as determined on the SP142 PD-L1 immunohistochemistry assay, with positivity defined as immune cells greater than or equal to (>/=) 1%
* Spinal cord compression not definitively treated with surgery and/or radiation or previously diagnosed and treated spinal cord compression without evidence that disease has been clinically stable for >2 weeks prior to initiation of study treatment
* Known central nervous system (CNS) disease, except for treated asymptomatic CNS metastases
* Leptomeningeal disease

Cohort B:

* History of invasive breast cancer
* Stage IV (metastatic) breast cancer
* Prior systemic therapy for treatment and prevention of breast cancer
* Previous therapy with anthracyclines, platinum, or taxanes for any malignancy
* Synchronous, bilateral invasive breast cancer
* Cardiopulmonary dysfunction

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 83 (Actual)
Dates: Start 2020-09-28 (Actual); Primary Completion 2023-03-08 (Actual); Study Completion 2023-03-08 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants With Adverse Events (Cohort B) | Up to approximately 21 months
Confirmed Objective Response Rate ORR (Cohort A) | Up to approximately 21 months

SECONDARY OUTCOMES:
Percentage of Participants With Adverse Events (Cohort A) | Up to approximately 21 months
Progression-free Survival (Cohort A) | Up to approximately 21 months
Duration of Response (Cohort A) | Up to approximately 21 months
Overall Survival (Cohort A) | Up to approximately 21 months
Serum Concentrations of Tiragolumab | Cohort A: Day 1 of Cycles (cycle=28 days) 1, 2, 3, 4, 8, 12, and 16 and at TD visit from start of treatment up to approximately 17 months; Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
  TD visit: treatment discontinuation visit
Serum Concentrations of Atezolizumab | Cohort A: Day 1 of Cycles (cycle=28 days) 1, 2, 3, 4, 8, 12, and 16 and at TD visit from start of treatment up to approximately 17 months; Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Plasma Concentrations of Nab-paclitaxel (Cohort B) | Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Plasma Concentrations of Carboplatin (Cohort B) | Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Plasma Concentrations of Doxorubicin (Cohort B) | Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Plasma Concentrations of Cyclophosphamide (Cohort B) | Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Percentage of Participants With Anti-drug Antibodies (ADAs) to Tiragolumab | Cohort A: Day 1 of Cycles (cycle=28 days) 1, 2, 3, 4, 8, 12, and 16 and at TD visit from start of treatment up to approximately 17 months; Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months
Percentage of Participants With ADAs to Atezolizumab | Cohort A: Day 1 of Cycles (cycle=28 days) 1, 2, 3, 4, 8, 12, and 16 and at TD visit from start of treatment up to approximately 17 months; Cohort B: Day 1 of Cycles (cycle=28 days) 1-5 and at TD visit from start of treatment up to approximately 5 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trial, Study Director — Hoffmann-La Roche
Locations (24):
- United States (5):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Univ of Chicago, Chicago, Illinois
  - Levine Cancer Institute, Charlotte, North Carolina
  - Magee-Woman's Hospital, Pittsburgh, Pennsylvania
  - Tennessee Onc., PLLC - SCRI, Nashville, Tennessee
- Australia (2):
  - Mater Hospital; Cancer Services, South Brisbane, Queensland
  - Fiona Stanley Hospital; FSH Cancer Centre Clinical Trials Unit, Bull Creek, Western Australia
- Brazil (4):
  - Hospital Sao Rafael - HSR, Salvador, Estado de Bahia
  - Hospital Araujo Jorge; Departamento de Ginecologia E Mama, Goiânia, Goiás
  - Hospital Sírio-Libanês, São Paulo, São Paulo
  - Clinica de Pesquisa e Centro de Estudos em Oncologia Ginecologica e Mamaria Ltda, São Paulo, São Paulo
- Germany (2):
  - Klinikum Essen-Mitte Ev. Huyssens-Stiftung / Knappschafts GmbH; Klinik für Senologie / Brustzentrum, Essen
  - Nationales Centrum für Tumorerkrankungen (NCT) ; Gyn. Onk. Frauenklinik; Uniklinikum Heidelberg, Heidelberg
- Russia (3):
  - Arkhangelsk Regional Clinical Oncology Dispensary, Arkhangelsk, Arhangelsk
  - SBIH "Moscow Clinical Scientific and Practical Center named after A.S. Loginov of DHM", Moskva, Moscow Oblast
  - Blokhin Cancer Research Center; Combined Treatment, Moskva, Moscow Oblast
- South Korea (3):
  - Severance Hospital, Yonsei University Health System, Seoul
  - Seoul National University Hospital, Seoul
  - Asan Medical Center, Seoul
- Spain (3):
  - Complejo Hospitalario Universitario de Santiago (CHUS) ; Servicio de Oncologia, Santiago de Compostela, LA Coruña
  - Hospital Universitario Virgen Macarena; Servicio de Oncologia, Seville
  - Hospital Clínico Universitario de Valencia; Servicio de Oncología, Valencia
- Taiwan (2):
  - China Medical University Hospital; Surgery, Taichung
  - National Taiwan Uni Hospital; General Surgery, Taipei

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to individual patient level data through the clinical study data request platform (www.vivli.org). Further details on Roche's criteria for eligible studies are available here (https://vivli.org/ourmember/roche/). For further details on Roche's Global Policy on the Sharing of Clinical Information and how to request access to related clinical study documents, see here (https://www.roche.com/research_and_development/who_we_are_how_we_work/clinical_trials/our_commitment_to_data_sharing.htm).

REFERENCES:
- [Derived] Kuemmel S, Jung KH, Andrade L, Assad-Suzuki D, de la Cruz Merino L, Freitas-Junior R, Hegg R, Huang CS, Martin H, Schneeweiss A, Dieterich M, Nguyen Duc A, Feng Y, Meng R, Swat A, Seiller A, Bermejo B, Hamilton EP. Safety and efficacy of tiragolumab, atezolizumab and chemotherapy for early-stage or PD-L1-positive advanced triple-negative breast cancer: a phase Ib study. ESMO Open. 2025 Dec;10(12):105869. doi: 10.1016/j.esmoop.2025.105869. Epub 2025 Nov 25. PMID 41297162